CLINICAL TRIAL: NCT00828776
Title: Clinical Trial of Pharmacodynamic Effects and Non-Clinical Inferiority of the Drug Heparin Sodium Produced by the Laboratory Cristália When Compared With the Product Liquemine of Roche Laboratory in Patients With Chronic Renal Failure
Brief Title: Pharmacodynamics and Non-Clinical Inferiority of Heparin Sodium (Cristália) Compared With the Product Liquemine (Roche) in Chronic Renal Failure
Acronym: heparin
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEPCRI0907
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2009-01-26 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Renal Failure
Keywords: TTPa; Anti-Xa; Adverse Reactions
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Heparin Cristália
  Interventions: Biological: Heparin sodic - Cristália
- 2 (Active Comparator): Heparin - Roche
  Interventions: Biological: heparin - Liquemine (Roche)

INTERVENTIONS:
Biological: Heparin sodic - Cristália — 5000UI/mL
  Arms: 1
Biological: heparin - Liquemine (Roche) — 5000UI/mL
  Arms: 2

SUMMARY:
The primary objective of the study was to assess the safety in use of the drug Heparin Sodium, produced by Cristália Laboratory, compared drug Liquemine ®, manufactured by Roche Laboratory, and secondary purpose was to evaluate the non-inferiority clinical testing of the product on the product comparator and pharmacodynamic effect, as evidenced by analyzing the parameters and TTPA Anti-Xa in patients with chronic renal failure in treatment of hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes, regardless of color or social class
* Age over 18 years with a good clinical medical criteria
* Patients who agreed to participate and signed the Informed Consent
* Insufficient patients in chronic renal dialysis schedule (3 times per week)
* Patients with creatinine clearance <30ml/min
* Patients with indication for anticoagulation during hemodialysis

Exclusion Criteria:

* Patients with sensitivity to heparin sodium;
* Patients with hypersensitivity to benzyl alcohol
* Patients with a history of bleeding or illness that can change the blood coagulation aggravate or terminate the clinical picture, such as tables of gastric ulcer
* Patients with a history of peptic ulcer
* Patients with body mass index greater than 30
* Cancer patients because of the possibility of compromising the function of the variable coagulation
* Patients in period of pregnancy or after delivery
* Patients with genetic abnormality of the clotting system
* Polytraumatized patients
* Patients using glucocorticoids for at least 1 month
* Patients using other anticoagulants
* Patients with high rate of bleeding
* Patients undergoing any surgery performed less than 15 days due to the risk of training of hematoma at the site of surgery
* Hypertension above 140/90 mmHg
* Patients using medications that could affect hemostasis
* Patients using the following medicines: hormonal anti not including Ketorolac; Dextran 40, ticlopidine and clopidogrel, systemic glucocorticoids, thrombolytic agents and anticoagulants and other antiplatelet agents, including antagonists of glycoprotein IIb / IIIa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
TTPA Anti-Xa Adverse Reactions | 12 consecutive sessions of hemodialysis

CONTACTS AND LOCATIONS:
Locations (1):
- Lal Clinica Pesquisa E Desenvolvimento Ltda, Valinhos, São Paulo, Brazil